CLINICAL TRIAL: NCT03227614
Title: Friends/Family in the Abortion Procedure Room (FAIR): Assessing Pain Level, Patient, Staff and Support Person Satisfaction With Support Person in Abortion Procedure Room: A Randomized Controlled Trial
Brief Title: Friends/Family in the Abortion Procedure Room (FAIR)
Acronym: FAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Planned Parenthood of Southwest and Central Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00019968
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Anxiety; Pain; Abortion
Keywords: abortion; social support; Anxiety; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This arm of participants will not experience the intervention of having a support person of the patient's choice support the patient during their abortion.
- Support Person Intervention (Experimental): This arm of participants will experience the intervention of having a support person of the patient's choice support them during their abortion procedure.
  Interventions: Behavioral: Support Person Intervention

INTERVENTIONS:
Behavioral: Support Person Intervention — The patient participant will have a support person of her choice accompany her during her abortion procedure.
  Arms: Support Person Intervention

SUMMARY:
This study aims to explore patient, support person, and health care providers' experience and satisfaction with social support in the abortion procedure room. Although some providers do allow a support person in the abortion procedure room, no study has formally examined the effects of this practice.

If this study demonstrates higher patient satisfaction and lower perceptions of pain and anxiety levels in patients who have social support in the in-clinic abortion procedure room, this could change standard procedures in the in-clinic abortion procedure room, allowing for more positive patient experiences.

DETAILED DESCRIPTION:
Having an abortion is a complexly emotional experience for many women. Women with strong social support, from a partner, friend or family member, report better psychological adjustment. During medication abortion, patients reported high satisfaction levels, in part, because of being able to share the experience with another person. During in-clinic abortion, patients report lower levels of anxiety when they have a support person (partner, spouse, friend or family member) in the post-abortion recovery room. Additionally, support persons indicate feeling they can successfully comfort the woman. In the abortion procedure room, doula support has a positive psychological impact on patients and decreases the need for additional clinic support resources. Because doula support in the abortion procedure room and social support in the post-abortion recovery room improves patient experience, it is reasonable to believe that having a support person in the procedure room may also improve patient experience. However, there are no data about the patient, support person, and health care provider's experience and satisfaction with a support person in the abortion procedure room.

This study aims to explore patient, support person, and health care providers' experience and satisfaction with social support in the abortion procedure room. Although some providers do allow a support person in the abortion procedure room, no study has formally examined the effects of this practice.

If this study demonstrates higher patient satisfaction and lower perceptions of pain and anxiety levels in patients who have social support in the in-clinic abortion procedure room, this could change standard procedures in the in-clinic abortion procedure room, allowing for more positive patient experiences.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Any patient who presents and consents for dilation and curettage
* Patient participants 17 and younger must have a legal guardian provide consent for participation, and the patient must provide assent
* Ability to provide written informed consent in English and comply with all study procedures

Support Persons:

* Any person 18 years and older who the patient selects to accompany as their support person
* Ability to provide written informed consent in English and comply with all study procedures

Health Care Providers:

* Any health center staff attending to the enrolled patient in both intervention and control arms of the study
* Ability to provide written informed consent in English and comply with all study procedures

Exclusion Criteria:

* Patients without a support person on-site willing to participate
* Patients or support persons that are unable to provide written informed consent in English and comply with all study procedures.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
Anxiety | 1 day
  Evaluating anxiety through State Trait Anxiety Inventory (STAI)

SECONDARY OUTCOMES:
Perceived Pain | 1 day
  Patient Subject will take VAS Pain Scale to evaluate perceived pain

CONTACTS AND LOCATIONS:
Locations (1):
- Planned Parentehood of Southwest and Central Florida (PPSWCF), Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Major B, Cozzarelli C, Sciacchitano AM, Cooper ML, Testa M, Mueller PM. Perceived social support, self-efficacy, and adjustment to abortion. J Pers Soc Psychol. 1990 Sep;59(3):452-63. doi: 10.1037//0022-3514.59.3.452. PMID 2231279
- [Background] Kero A, Lalos A, Hogberg U, Jacobsson L. The male partner involved in legal abortion. Hum Reprod. 1999 Oct;14(10):2669-75. doi: 10.1093/humrep/14.10.2669. PMID 10528006
- [Background] Kero A, Lalos A. Reactions and reflections in men, 4 and 12 months post-abortion. J Psychosom Obstet Gynaecol. 2004 Jun;25(2):135-43. doi: 10.1080/01674820400000463. PMID 15715036
- [Background] Kero A, Lalos A, Wulff M. Home abortion - experiences of male involvement. Eur J Contracept Reprod Health Care. 2010 Aug;15(4):264-70. doi: 10.3109/13625187.2010.485257. PMID 20809674
- [Background] Veiga MB, Lam M, Gemeinhardt C, Houlihan E, Fitzsimmons BP, Hodgson ZG. Social support in the post-abortion recovery room: evidence from patients, support persons and nurses in a Vancouver clinic. Contraception. 2011 Mar;83(3):268-73. doi: 10.1016/j.contraception.2010.07.019. Epub 2010 Sep 15. PMID 21310290
- [Background] Chor J, Hill B, Martins S, Mistretta S, Patel A, Gilliam M. Doula support during first-trimester surgical abortion: a randomized controlled trial. Am J Obstet Gynecol. 2015 Jan;212(1):45.e1-6. doi: 10.1016/j.ajog.2014.06.052. Epub 2014 Jun 28. PMID 24983679
- [Background] Krohne HW, Slangen KE. Influence of social support on adaptation to surgery. Health Psychol. 2005 Jan;24(1):101-5. doi: 10.1037/0278-6133.24.1.101. PMID 15631568
- [Background] Jensen MP, Miller L, Fisher LD. Assessment of pain during medical procedures: a comparison of three scales. Clin J Pain. 1998 Dec;14(4):343-9. doi: 10.1097/00002508-199812000-00012. PMID 9874014

DOCUMENTS (2):
  • Study Protocol (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT03227614/Prot_000.pdf
  • Informed Consent Form (2017-04-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT03227614/ICF_001.pdf